CLINICAL TRIAL: NCT03015688
Title: the New Biomarker of the Knee Osteoarthritis Knee Osteoarthritis Occurrence and Progression
Status: Completed | Type: Observational
Sponsor: Shihezi University (Other)
Responsible Party: Principal Investigator, Jianwei He, Principal investigator, Shihezi University
Other Study IDs: 2012-06-01
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Knee Osteoarthritis
Keywords: Biomarkers
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

GROUPS / COHORTS (2):
- knee OA: OA diagnosis was on the basis of the diagnosis and treatment guideline of the American Academy of Orthopedic Surgeons Participants who met the following criteria were excluded：the knee OA concomitant with hip OA, suppurative and rheumatoid arthritis, gout patients, patients who underwent knee arthroscopy surgery within 6 months, bilateral or unilateral knee replacements, the knee joint trauma patients, histories of glucocorticoid and/or sterol hormones.
  Interventions: Radiation: x-ray images
- Control: "no often have pain, aching or stiffness in your Left/right knee during last month","no Left/right knee trauma history","no histories of glucocorticoid and/or sterol hormones" normal knee X-ray images,
  Interventions: Radiation: x-ray images

INTERVENTIONS:
Radiation: x-ray images

SUMMARY:
It was previously proved an association of TGF-β1 and PDGF-BB with the pathogenesis of osteoarthritis (OA) by experiments of OA animal models. In this study, we aimed to determine whether serum concentrations of TGF-β1, PDGF-BB and CTX-1 were related to the knee OA. knee OA cases were collected from the first affiliated hospital of Shihezi university and healthy controls were recruited from the community. The severity of knee OA was defined as kellgren-lawrence (K-L) classification criteria.Serum levels of chemical biomarkers were compared between knee OA cases and controls or among K-L grade 2 to grade 4 groups. The serum concentrations of the TGF-β1, PDGF-BB and CTX-1 were determined by ELISA .

ELIGIBILITY:
Inclusion Criteria:

* OA diagnosis was on the basis of the diagnosis and treatment guideline of the American Academy of Orthopedic Surgeons

Exclusion Criteria:

Participants who met the following criteria were excluded：

* the knee OA concomitant with hip OA,
* suppurative and rheumatoid arthritis,
* gout patients,
* patients who underwent knee arthroscopy surgery within 6 months,
* bilateral or unilateral knee replacements,
* the knee joint trauma patients,
* histories of glucocorticoid and/or sterol hormones.

Ages: 38 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 210 patients diagnosed with knee OA in clinics were found in hospital patients .
  Healthy controls were recruited from community questionnaires in Shihezi city, Xinjiang province, China.
Sampling Method: Probability Sample
Enrollment: 460 (Actual)
Dates: Start 2012-06; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Serum levels of Transforming Growth Factor Beta1 (TGF-β1) and Platelet Derived Growth Factor BB (PDGF-BB) may be novel biomarkers in knee osteoarthritis | 3 years